CLINICAL TRIAL: NCT05708287
Title: The Physiologic Effect of the Flow Generated by High Flow Nasal Cannula in Mild Respiratory Failure a Prospective Study
Brief Title: The Physiologic Effect of the Flow Generated by High Flow Nasal Cannula in Mild Respiratory Failure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: HMO-20-0260
Record Dates: First submitted 2022-12-14; First posted 2023-02-01 (Actual); Last update posted 2023-02-01 (Actual); Status verified 2022-12

CONDITIONS: Respiratory Failure
Keywords: high flow nasal cannula; oxygenation; ventilation; conventional oxygen therapy; Arterial Blood Gasses
MeSH Terms: conditions — Respiratory Insufficiency; Respiratory Aspiration

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- all patients (Experimental)
  Interventions: Device: HFNC

INTERVENTIONS:
Device: HFNC — The patients with mild hypoxemia, defined as the need for conventional oxygen therapy (COT) using nasal cannula at 4-5 liters per minute (LPM) to maintain O2 Saturation >90%, were commenced on HFNC therapy

SUMMARY:
High flow nasal cannula (HFNC) oxygen therapy is increasingly used for hypoxemic respiratory failure and is proving useful in avoiding or delaying intubation and mechanical ventilation. However, basic information regarding the physiologic effects of this method is missing. In this study, the effects of oxygen delivery by HFNC on oxygenation, ventilation and cardiovascular vital signs in patients with mild hypoxemic respiratory failure were evaluated.

DETAILED DESCRIPTION:
Oxygen (O2) therapy delivered by means of High Flow Nasal Cannula (HFNC) is being increasingly used. This device, capable of delivering high flow, oxygen enriched gas, has been shown to reduce intubation rates in patients with hypoxemic respiratory failure. The primary components of HFNC are "nasal prongs" (or cannulae) that are inserted into the nostrils, a device which provides a warmed and humidified air / oxygen mixture and regulators that control oxygen concentration, temperature and total gas flow. Commercially available systems can deliver up to 40 - 60 liters per minute (LPM) of oxygen flow.

This method of non-invasive oxygen delivery has several presumed important working principals. Firstly, the high flow rate may meet the patient's own inspiratory flow rate. This enables accurate delivery of a high fractional inspired concentration of oxygen (FiO2). Second, the high gas flow might also produce a certain degree of Continuous Positive Airway Pressure (CPAP). In addition, the heated and humidified gas might also wash out/reduce the physiological airway dead space of the patient. Furthermore, HFNC is more comfortable and might be better tolerated than other Non-Invasive Ventilation (NIV) devices, such as Bi-level positive airway pressure (BiPAP). This, in turn, can prolong the time the patient is comfortably connected to the HFNC device.

Information regarding the basic physiologic influence of HFNC on oxygenation, ventilation and vital signs is missing in the literature. Patients with mild respiratory failure provide an opportunity to examine this topic. On one hand, these patients suffer from respiratory failure manifested by hypoxemia, on the other hand the respiratory failure is mild to the extent that removal of the conventional oxygen therapy (COT) will not lead to immediate respiratory collapse. This prospective study evaluates the physiologic effects of HFNC in 28 patients with mild respiratory failure.

ELIGIBILITY:
Inclusion Criteria:

* Minimal age 18
* The patient had invasive blood pressure monitoring via an arterial line in situ
* The patient had a mild respiratory failure manifested by the need for oxygen support via nasal prongs in order to maintain oxygen saturation (SpO2) above 90% for at least one hour prior to the start of the intervention

Exclusion Criteria:

* Shortness of breath
* Patients regularly using O2 at home
* No patient consent for participation

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2020-08-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
The effect of changing flow rates generated by HFNC on oxygenation parameters of 28 patients with mild respiratory failure | 60 minutes
  Change in PaO2 in mmHg(Partial pressure of oxygen in arterial blood) from baseline on nasal cannula and after giving gradually increasing flow rates to 60 Liters Per Minute on HFNC, at constant FiO2 of 40%.
The effect of changing flow rates generated by HFNC on ventilation parameters of 28 patients with mild respiratory failure | 60 minutes
  Change in PaCO2 in mmHg(Partial pressure of carbon dioxide in arterial blood) from baseline on nasal cannula and after giving gradually increasing flow rates to 60 Liters Per Minute on HFNC, at constant FiO2 of 40%.

CONTACTS AND LOCATIONS:
Locations (1):
- Hadassah medical center, Jerusalem, Israel